CLINICAL TRIAL: NCT06276608
Title: Iron Deficiency in Pediatric Heart Surgery: Impact on Anemia, Transfusion and Complications, a Retrospective Cohort Study
Brief Title: Iron Deficiency in Pediatric Heart Surgery
Status: Recruiting | Type: Observational
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PED_Fe_def
Record Dates: First submitted 2024-02-13; First posted 2024-02-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Iron Deficiencies; Iron Deficiency Anemia; Cardiac Surgical Procedures; Congenital Heart Disease in Children
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric cardiac surgery patients: All patients who underwent pediatric cardiac surgery in our institution between January 1, 2019 and december 31, 2023
  Interventions: Diagnostic Test: Iron status

INTERVENTIONS:
Diagnostic Test: Iron status — Iron status will be based on preoperative ferritin levels: a ferritin < 10 mcg/L will be considered as iron deficiency, ferritin levels > 10 mcg/L will be considered normal

SUMMARY:
The prevalence of iron deficiency in pediatric cardiac surgery patients is not very well known. Iron deficiency can lead to anemia, higher transfusion rates and possibly higher complication rates. In this retrospective study, the iron status of all patients undergoing pediatric cardiac surgery at our institution between January 2019 and december 2023 will be analyzed. Together with iron status, transfusion requirements as well as complications will be recorded. Iron status will be reported with descriptive statistics, patients with or without iron deficiency will be compared using non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent pediatric cardiac surgery at our institution between January 1, 2019 and December 31, 2023

Exclusion Criteria:

* Incomplete medical charts
* Patients who did not consent to the use of their medical data

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: All patients who underwent pediatric cardiac surgery at our institution between January 1, 2019 and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of preoperative iron deficiency (%) | 24 hours
  A preoperative ferritin < 10 mcg/L will be considered as iron deficiency. Iron deficiency will be reported using descriptive statistics (mean, standard deviation, median, interquartile range, %)
Complications | 28 days
  The complication rate (%) will be reported. Complications are defined by the occurence of one or more of the following events:
  * transfusion rate (%)
  * volume of packed red cells transfused (mL/kg)
  * perioperative blood loss (mL/kg)
  * need for surgical re-exploration (%)
  * intensive care stay (days)
  * new renal insufficiency (%)
  * use of inotropes (%)
  * 28 day mortality (%) The frequency of any single item will also be reported (%)

CONTACTS AND LOCATIONS:
Locations (1):
- H.U.B - Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao P, Wang X, Zhang P, Jin Y, Bai L, Wang W, Li Y, Liu J. Preoperative Iron Deficiency Is Associated With Increased Blood Transfusion in Infants Undergoing Cardiac Surgery. Front Cardiovasc Med. 2022 Jun 2;9:887535. doi: 10.3389/fcvm.2022.887535. eCollection 2022. PMID 35722123
- [Background] Sidhu S, Kakkar S, Dewan P, Bansal N, Sobti PC. Adherence to Iron Chelation Therapy and Its Determinants. Int J Hematol Oncol Stem Cell Res. 2021 Jan 1;15(1):27-34. doi: 10.18502/ijhoscr.v15i1.5247. PMID 33613898
- [Background] Temel HH, Kumbasar U, Buber E, Aksoy Y, Cavdar S, Dogan R, Demircin M, Pasaoglu I. Comparison of antioxidant reserve capacity of children with acyanotic & cyanotic congenital heart disease. Indian J Med Res. 2020 Dec;152(6):626-632. doi: 10.4103/ijmr.IJMR_2215_18. PMID 34145102
- [Background] Christen S, Finckh B, Lykkesfeldt J, Gessler P, Frese-Schaper M, Nielsen P, Schmid ER, Schmitt B. Oxidative stress precedes peak systemic inflammatory response in pediatric patients undergoing cardiopulmonary bypass operation. Free Radic Biol Med. 2005 May 15;38(10):1323-32. doi: 10.1016/j.freeradbiomed.2005.01.016. PMID 15855050